## Sangamo BioSciences, Inc.

## Clinical Approval Signature Page

**Protocol Number:** 

SB-728mR-1401

**Protocol Title:** 

A Phase 1/2 Open-Label Study to Assess the Safety and Tolerability of

Repeat Doses of Autologous T-Cells Genetically Modified at the CCR5 Gene by Zinc Finger Nucleases in HIV-Infected Subjects

Following Cyclophosphamide Conditioning

**Amendment 2:** 

October 10, 2014

Winson Tang, M.D.

Vice President, Clinical Research

Date

10/14/11/ Date

Dale Ando, M.D.

Vice President Therapeutic Development and CMO